CLINICAL TRIAL: NCT05821868
Title: Contrasting Dosivent Spacer Device With Plus Flow Vu Spacer in Bronchial Hyperreactivity Participants
Brief Title: Contrasting Dosivent With Plus Flow Vu Spacer in Bronchial Hyperreactivity Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Luis Puente Maestu, Principal Investigator, Hospital General Universitario Gregorio Marañon
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 001
Record Dates: First submitted 2023-02-22; First posted 2023-04-20 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Bronchial Hyperreactivity; Inhalant Use
MeSH Terms: conditions — Bronchial Hyperreactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerochamber Plus® Flow-Vu® (Active Comparator): 1. Inhaled space chamber commonly use in our lung function lab for Bronchodilator Testing
  Interventions: Device: Aerochamber Plus Flow Vu
- Dosivent (Experimental): 2. Newer and different inhaled space chamber for Bronchodilator Testing
  Interventions: Device: Dosivent

INTERVENTIONS:
Device: Dosivent — Dosivent® inhalation chamber is designed to optimize the delivery of inhaled bronchodilators and corticosteroids in the treatment of respiratory diseases
  Arms: Dosivent
Device: Aerochamber Plus Flow Vu — Aerochamber Plus Flow Vu® inhalation chamber is also designed to optimize the delivery of inhaled bronchodilators and corticosteroids in the treatment of respiratory diseases
  Arms: Aerochamber Plus® Flow-Vu®

SUMMARY:
This study aims to compare the efficacy, as measured by changes in forced expiratory volume in the first second (FEV1) and forced vital capacity (FVC), of salbutamol inhaled with the Dosivent® chamber versus the widely used Aerochamber Plus® Flow-Vu® in participants with a positive bronchodilator testing.

DETAILED DESCRIPTION:
The investigators are conducting a non-randomized, open-label, crossover-controlled clinical trial in 50 participants with a previous positive bronchodilation testing. The protocol was approved by the local clinical ethics committee (code 03/2022). All participants provided written informed consent before any study procedure. During the study, the principles of the Declaration of Helsinki and the current standards of Good Clinical Practice were followed.

Participants over 18 years of age are included who attended our center for a bronchodilator test, gave a positive result in this test, and provided written informed consent for participation in this study. Participants are excluded if grade A quality spirometry was not obtained according to the classification in current regulations and, in the opinion of the investigator, performing a bronchodilator test could pose a risk to the participant or interrupting the usual bronchodilator treatment could worsen the underlying respiratory pathology.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years of age
* Attending our center for a bronchodilator test
* Positive bronchodilator result with increase of Forced Expiratory Volume in first second greater than 200 mililiters and 12%
* Provided written informed consent for participation in this study

Exclusion Criteria:

* Grade A quality spirometry was not obtained according to the classification in current regulation
* Performing a bronchodilator test, in the opinion of the investigator, could pose a risk to the participant or interrupting the usual bronchodilator treatment could worsen the underlying respiratory pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of bronchodilator response in forced expiratory volume in the first second (FEV1) in miliLiters between Dosivent® and Aerochamber Plus® Flow-Vu® chambers in participants with bronchial hyperreactivity | 12 months
  This study aim is to compare the efficacy, as measured by changes in forced expiratory volume in the first second (FEV1) in mililiters of inhaled Salbutamol with the Dosivent® chamber versus the widely used Aerochamber Plus® Flow-Vu® in participants with a positive Bronchodilator testing.
Comparison of bronchodilator response in forced expiratory volume in the first second (FEV1) in percentage between Dosivent® and Aerochamber Plus® Flow-Vu® chambers in participants with bronchial hyperreactivity | 12 months
  This study aim is to compare the efficacy, as measured by changes in forced expiratory volume in the first second (FEV1) in percentage of inhaled salbutamol with the Dosivent® chamber versus the widely used Aerochamber Plus® Flow-Vu® in participants with a positive Bronchodilator testing.

SECONDARY OUTCOMES:
Comparison of bronchodilator response forced vital capacity (FVC) in miliLiters between Dosivent® and Aerochamber Plus® Flow-Vu® chambers in participants with bronchial hyperreactivity | 12 months
  This study aim is to compare the efficacy, as measured by changes in forced vital capacity (FVC) in mililiters,of inhaled Salbutamol with the Dosivent® chamber versus the widely used Aerochamber Plus® Flow-Vu® in participants with a positive Bronchodilator testing.
Comparison of bronchodilator response forced vital capacity (FVC) in percentage between Dosivent® and Aerochamber Plus® Flow-Vu® chambers in participants with bronchial hyperreactivity | 12 months
  This study aim is to compare the efficacy, as measured by changes in forced vital capacity (FVC) in percentage,of inhaled Salbutamol with the Dosivent® chamber versus the widely used Aerochamber Plus® Flow-Vu® in participants with a positive Bronchodilator testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañon, Madrid, Spain

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05821868/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05821868/ICF_001.pdf